CLINICAL TRIAL: NCT03668340
Title: A Phase 2 Study of the Wee1 Inhibitor AZD1775 in Women With Recurrent or Persistent Uterine Serous Carcinoma or Uterine Carcinosarcoma
Brief Title: AZD1775 in Women With Recurrent or Persistent Uterine Serous Carcinoma or Uterine Carcinosarcoma
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Principal Investigator, Joyce Liu, MD, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 18-316
Record Dates: First submitted 2018-09-11; First posted 2018-09-12 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Uterine Cancer
Keywords: Uterine Cancer
MeSH Terms: conditions — Uterine Neoplasms | interventions — adavosertib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Part A: AZD1775 (Experimental): -AZD1775 will be taken by mouth daily on days 1 through 5 and days 8 through 12 of each 21-day cycle
  Interventions: Drug: AZD1775
- Part B: AZD1775 in Carcinosarcoma (Experimental): -AZD1775 will be taken by mouth daily on days 1 through 5 and days 8 through 12 of each 21-day cycle
  Interventions: Drug: AZD1775
- Part C: AZD1775 in Uterine Serous with biopsiable disease (Experimental): -AZD1775 will be taken by mouth daily on days 1 through 5 and days 8 through 12 of each 21-day cycle
  Interventions: Drug: AZD1775

INTERVENTIONS:
Drug: AZD1775 — AZD1775 blocks the activity of Wee1, a protein that helps to regulate how cells divide and grow. Certain cancer cells may be more vulnerable to having this process blocked

SUMMARY:
This research study is studying an investigational drug as a possible treatment for uterine cancer.

The drug involved in this study is:

-AZD1775

DETAILED DESCRIPTION:
This research study is a Phase II clinical trial. Phase II clinical trials test the safety and effectiveness of an investigational drug to learn whether the drug works in treating a specific disease. "Investigational" means that the drug is being studied.

The FDA (the U.S. Food and Drug Administration) has not approved AZD1775 as a treatment for any disease.

The "investigational drug" AZD1775 is being given alone to patients with this type of cancer. AZD1775 is also being studied in lung cancer, ovarian cancer, and other solid tumors throughout the world. AZD1775 blocks the activity of Wee1, a protein that helps to regulate how cells divide and grow. Certain cancer cells may be more vulnerable to having this process blocked. This study is being done to assess the safety and effectiveness of AZD1775 to learn if AZD1775 works in treating this type of cancer.

ELIGIBILITY:
Inclusion Criteria:

* Participants in Parts A and C must have histologically or cytologically confirmed recurrent or persistent uterine serous carcinoma. For the purposes of this study, uterine carcinomas (with the exception of carcinosarcomas) that have any component that is considered serous will be considered a uterine serous carcinoma.
* Participants in Part B must have histologically or cytologically confirmed recurrent uterine carcinosarcoma. Additionally, the following features must also be present:

  * Presence of a p53 alteration (by either IHC or next generation sequencing)
  * Metastatic or extra-uterine component must be confirmed on pathology to be from the carcinoma component of the disease
  * Patients without confirmation that the metastatic or extrauterine component of disease is of carcinoma histology may be considered after discussion with the PI
* Participants must have measurable disease, defined as at least one lesion that can be accurately measured per RECIST 1.1 criteria. See Section 11 for the evaluation of measurable disease.
* Participants must have had one prior platinum-based chemotherapy regimen for management of advanced or metastatic uterine serous carcinoma or uterine carcinosarcoma. Chemotherapy administered only in conjunction with primary RT as a radiosensitizer should not count as a systemic regimen. There is no restriction on the number of prior lines of therapy a participant may have previously received.
* Age 18 years or older.
* ECOG performance status 0 or 1 (see Appendix A)
* Participants must have normal organ and marrow function as defined below:

  * absolute neutrophil count ≥1,500/mcL
  * hemoglobin ≥9 g/dL
  * platelets ≥100,000/mcL
  * total bilirubin ≤ upper limit of normal (ULN) or ≤1.5x ULN in patients with liver metastases or well-documented Gilbert's Syndrome.
  * AST(SGOT)/ALT(SGPT) ≤3 × ULN or ≤5 × ULN in patients with liver metastases
  * creatinine ≤1.5 × ULN OR
  * creatinine clearance ≥45 mL/min/1.73 m2 as calculated by the Cockroft-Gault method for participants with creatinine levels above institutional normal.
* Willingness to release archival tissue for research purposes.
* Participants in Part C must have biopsiable disease (in a lesion that is not being utilized as the target lesion for RECIST assessment) and be willing to undergo pre- and on-treatment biopsies. Participants in Part B with biopsiable disease must be willing to undergo pre- and on-treatment biopsies.
* The effects of AZD1775 on the developing human fetus are unknown. For this reason, women of child-bearing potential must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) from 2 weeks prior to study entry and for 1 month after study drug discontinuation. Please see Appendix C for "Definition Women of Childbearing Potential and Acceptable Contraceptive Methods." Patients of child-bearing potential should not be breastfeeding, and must have a negative serum or urine pregnancy test within 3 days prior to the start of study treatment. Should a woman become pregnant or suspect she is pregnant while she is participating in this study, she should inform her treating physician immediately.
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Participants who have had chemotherapy, radiotherapy, or investigational therapy within 3 weeks (6 weeks for nitrosoureas or mitomycin C) prior to first dose of AZD1775, or those who have not recovered to Grade 1 from adverse events (excluding alopecia or anorexia) due to agents administered more than 3 weeks earlier. Participants may not have had hormonal therapy within 2 weeks of the first dose of AZD1775.
* Participants who are receiving any other investigational agents.
* Participants who have MSI-high or MMR-deficient tumors will not be eligible unless they have already received prior therapy with pembrolizumab or another PD1/PD-L1 immune checkpoint inhibitor or are deemed not to be a candidate for immune checkpoint therapy.
* Participants with known brain metastases or other CNS disease should be excluded from this clinical trial because of their poor prognosis and because they often develop progressive neurologic dysfunction that would confound the evaluation of neurologic and other adverse events. Participants with treated brain metastases that have no evidence of progression or hemorrhage for at least 2 weeks after treatment will be allowed on study.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to AZD1775.
* Participants may not have had prior receipt of a cell cycle checkpoint inhibitor (e.g., Chek1, Wee1, or ATR inhibition)
* Participants receiving any medications or substances that are sensitive CYP3A4 substrates or are CYP3A4 substrates with a narrow therapeutic index, or which are moderate to strong inhibitors/inducers of CYP3A4 which cannot be discontinued two weeks prior to Day 1 of dosing and withheld through the study until 2 weeks after the last dose of study drug. Co-administration of aprepitant or fosaprepitant during this study is prohibited.
* Transporter studies (in vitro) have shown that AZD1775 is an inhibitor of breast cancer resistance protein (BRCP). Please see Appendix B for additional details regarding prohibited drugs and drugs to be used with caution, including drugs affected by CYP3A4 or BRCP. Because the lists of these agents are constantly changing, it is important to also regularly consult a frequently-updated list such as http://medicine.iupui.edu/clinpharm/ddis/table.aspx; medical reference texts such as the Physicians' Desk Reference may also provide this information.
* Participants must not have undergone major surgical procedures within 28 days of beginning study treatment or minor surgical procedures within 7 days of beginning study treatment. Port-a-cath placement will be allowed within a 7 day window of starting study treatment.
* Participants must be able to swallow oral medication and may not have a percutaneous endoscopic gastrostomy (PEG) tube, be receiving total parenteral nutrition (TPN), or be dependent on IV fluid support.
* Participants with any of the following cardiac diseases currently or within the last 6 months as defined by the New York Heart Association (NYHA) ≥ Class 2 will not be eligible:

  * Unstable angina pectoris
  * Congestive heart failure
  * Acute myocardial infarction
  * Conduction abnormality not controlled with pacemaker or medication
  * Significant ventricular or supraventricular arrhythmias (patients with chronic rate-controlled atrial fibrillation in the absence of other cardiac abnormalities are eligible).
* Participants with a mean resting corrected QT interval (QTc) ≥ 480msec at study entry, as calculated by the Frederica formula (QTcF) by institutional standards obtained from an electrocardiogram (ECG) or congenital long QT syndrome. (Note: if one ECG demonstrates a QTcF >480 msec, then a mean QTcF of ≤ 480 msec obtained from 3 ECGs 2-5 minutes apart is required at study entry.
* Participants with any concomitant or prior invasive malignancies are ineligible with the following exceptions:

  * Treated limited-stage basal cell or squamous cell carcinoma of the skin
  * Carcinoma in situ of the breast or cervix
  * Prior cancer treated with curative intent with no evidence of recurrent disease 3 years following diagnosis and judged by the investigator to be at low risk of recurrence
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Pregnant women are excluded from this study because AZD1775 is an agent with an unknown potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with AZD1775, breastfeeding should be discontinued if the mother is treated with AZD1775.
* Known HIV-positive participants are ineligible because of the potential for pharmacokinetic interactions of antiretroviral medications with AZD1775 and the potential for an increased risk of lethal infections for these participants when treated with marrow-suppressive therapy.
* Because the composition, PK, and metabolism of many herbal supplements are unknown, the concurrent use of all herbal supplements is prohibited during the study (including, but not limited to, cannabis, St. John's wort, kava, ephedra [m huang], ginkgo biloba, dehydroepiandrosterone [DHEA], yohimbe, saw palmetto, and ginseng). Participants should stop herbal medications at least 7 days prior to first dose of AZD1775.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2018-10-22 (Actual); Primary Completion 2026-07-01 (Estimated); Study Completion 2027-07-01 (Estimated)

PRIMARY OUTCOMES:
Objective response rate | 2 years
  Response and progression will be evaluated in this study using the new international criteria proposed by the Response Evaluation Criteria in Solid Tumors (RECIST) guideline (version 1.1) [Eur J Ca 45:228-247, 2009]
Progression-free survival | 6 months
  Measured by the rate of progression-free survival at 6 months (PFS6) using RECIST v.1.1.

SECONDARY OUTCOMES:
Clinical benefit rate | 2 years
  Clinical benefit rate is defined as response rate plus stable disease x 6 months.
Duration of Response | 2 years
  The duration of overall response is measured from the time measurement criteria are met for CR or PR (whichever is first recorded) until the first date that recurrent or progressive disease is objectively documented.
Assess the toxicities of AZD1775 in women with recurrent or persistent uterine serous carcinoma or uterine carcinosarcoma using CTCAE v4 | 2 years
  Toxicities will be assessed using CTCAE v4.

CONTACTS AND LOCATIONS:
Overall Officials: Joyce Liu, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (1):
- Dana Farber Cancer Institute, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Liu JF, Xiong N, Campos SM, Wright AA, Krasner C, Schumer S, Horowitz N, Veneris J, Tayob N, Morrissey S, West G, Quinn R, Matulonis UA, Konstantinopoulos PA. Phase II Study of the WEE1 Inhibitor Adavosertib in Recurrent Uterine Serous Carcinoma. J Clin Oncol. 2021 May 10;39(14):1531-1539. doi: 10.1200/JCO.20.03167. Epub 2021 Mar 11. PMID 33705205